CLINICAL TRIAL: NCT03850106
Title: Effects of INDUS810 on Body Composition, Muscular Performance, and Training Adaptations During 12-weeks of Supplementation and Concurrent Training
Brief Title: Effects of INDUS810 on Body Composition, Muscular Performance, and Training Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Collaborators: Indus Biotech (Unknown)
Responsible Party: Principal Investigator, Jennifer Sandrock, Chief Operating Officer, The Center for Applied Health Sciences, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INDUS-PC-BC-2018
Record Dates: First submitted 2019-01-29; First posted 2019-02-21 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Weakness, Muscle
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (microcrystalline cellulose)
  Interventions: Dietary Supplement: Placebo
- Indus810 (Active Comparator): Indus810 ( 500mg/d)
  Interventions: Dietary Supplement: Indus810

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Indus810 — Active product
  Arms: Indus810

SUMMARY:
The purpose of this 12-week, interventional study is to determine the effects of oral supplementation with Indus810 (dietary supplement with active ingredient Fenugreek) on body composition, muscular performance, and training adaptations

DETAILED DESCRIPTION:
This 12-week study is a randomized, parallel-group, placebo-controlled, clinical trial of N=66 recreationally, but normal to moderately overweight/obese male subjects to be recruited at a single investigational center in Northeast Ohio (i.e. The Center for Applied Health Sciences).

Subjects will attend 4 study visits. At Visit 1, subjects will be screened for participation (i.e., medical history, physical exam, routine blood work, background baseline diet). At Visits 2 (day 0 - Baseline Testing), and 4 (week 12), measurements of various hemodynamic, hematologic & biochemical biomarkers of safety (Total testosterone, CBC, and comprehensive metabolic panel) will be made. At Visits 2, 3, and 4, the following efficacy measures will be obtained: Body Composition assessment via DEXA, Upper and Lower Body Performance testing on a Smith Machine and a TENDO unit utilizing the bench press and squat exercises, and anchored 100mm VAS scales (for various psychometric indices). In addition, a comprehensive side effect profile/ adverse event monitoring will take place throughout the 12-week study duration.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between the ages of 18 and 45.
* Body Mass Index (BMI):

  * 22-25; Waist:Hip Ratio 0.9-1
  * 25-35; Waist:Hip Ratio 0.85-1
* Normotensive (supine, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal supine, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, and fast for 8-10 hours prior each of the treatments.
* Has been participating in regular exercise training, at least 3 days per week, for the past 1-2 months.

Exclusion Criteria:

* History of diabetes.
* Use of any pre-workout or creatine containing products in the last 4 weeks.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic diseases that might impact absorption or amino acid metabolism, e.g. short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.). -Known sensitivity to any ingredient in the test formulations as listed in the Certificates- of-Analysis.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Concomitant use of corticosteroids or testosterone replacement therapy (ingestion, injection, or transdermal).
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Body composition | Change in score from Day 0 to day 56 and from day 0 to day 84
  body fat percentage (%)

SECONDARY OUTCOMES:
Upper body strength | Change in pounds from Day 0 to day 56 and from day 0 to day 84
  Weight lifted in pounds

CONTACTS AND LOCATIONS:
Overall Officials: Tim N Ziegenfuss, PhD, Principal Investigator — The Center for Applied Health Sciences
Locations (1):
- The Center for Applied Health Sciences, Stow, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided